CLINICAL TRIAL: NCT03593785
Title: A Phase I Randomized, Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD8233 Following Single Ascending Dose Administration to Healthy Male Subjects With Elevated LDL-C Levels.
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD8233 in Healthy Male Subjects With Increased Elevated LDL-C Levels.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D7990C00001
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Hypercholesterolemia
Keywords: Cholesterol; Biomarkers
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant
Masking Description: This study is single-blind with regard to treatment (AZD8233 or placebo) at each dose level.
  AZD8233 and placebo will be matched for formulation, appearance and amount. Subjects randomized to placebo will receive the same volume of injection as subjects on active drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): On Day 1, randomized subjects will receive single SC dose of AZD8233 dose 1 injection (6 subjects) or matching placebo (2 subjects).
  Interventions: Drug: AZD8233
- Cohort 2 (Experimental): On Day 1, randomized subjects will receive single SC dose of AZD8233 dose 2 injection (6 subjects) or matching placebo (2 subjects).
  Interventions: Drug: AZD8233
- Cohort 3 (Experimental): On Day 1, randomized subjects will receive single SC dose of AZD8233 dose 3 injection (6 subjects) or matching placebo (2 subjects).
  Interventions: Drug: AZD8233
- Cohort 4 (Experimental): On Day 1, randomized subjects will receive single SC dose of AZD8233 dose 4 injection (6 subjects) or matching placebo (2 subjects).
  Interventions: Drug: AZD8233
- Cohort 5 (Experimental): On Day 1, randomized subjects will receive single SC dose of AZD8233 dose 5 injection (6 subjects) or matching placebo (2 subjects).
  Interventions: Drug: AZD8233

INTERVENTIONS:
Drug: AZD8233 — Randomized subjects will receive single SC dose of AZD8233 (dose 1, dose 2, dose 3, dose 4 and dose 5) injection.

SUMMARY:
AZD8233 has not been evaluated in clinical studies previously. This is a first-in-human (FiH) study. This study will assess the safety, tolerability and pharmacokinetics (PK) of AZD8233, following subcutaneous (SC) administration of single ascending dose (SAD) of AZD8233. This study will also investigate the pharmacodynamics (PD) of AZD8233 by investigating the effect of AZD8233 on levels of cholesterol and related biomarkers.

DETAILED DESCRIPTION:
This randomized, single-blind, placebo-controlled study will be conducted at a single study center in United States of America. Up to 56 healthy male subjects with elevated LDL-C levels, aged 18 to 60 years will be randomized into this study. This study will consist of 5 cohorts with 8 subjects in each. Depending on emerging data, 2 additional cohorts may be added to test additional dose levels at the discretion of the sponsor, if the pre-defined exposure limits and stopping criteria have not been reached at previous administered doses. The study will comprise of 3 periods:

* A screening period of maximum 28 days.
* A treatment period:
* A follow-up period of 16 weeks

In each cohort, 6 subjects will be randomized to receive a single SC dose of AZD8233 and 2 subjects randomized to receive placebo. Single dose of AZD8233 SC injection (40 mg/mL) will be administered in each cohort as follows:

Cohort 1: Dose 1 (starting dose) Cohort 2: Dose 2 (provisional dose) Cohort 3: Dose 3 (provisional dose) Cohort 4: Dose 4 (provisional dose) Cohort 5: Dose 5 (provisional dose) Dosing for each ascending dose cohort will proceed with 2 subjects in a sentinel cohort, such that 1 subject will be randomized to receive placebo and 1 subject will be randomized to receive AZD8233.

In the treatment period, the sentinel and non-sentinel subjects will be resident at the clinical unit from the day before IMP administration (Day -1) until at least 72 hours and 48 hours after IMP administration, respectively.

Sentinel will have 10 follow-up visits (1, 2, 3, 4, 6, 8, 10, 12, 14 and 16 weeks post-dose). Non-sentinel subjects will have 11 follow-up visits (on Day 4 and 1, 2, 3, 4, 6, 8, 10, 12, 14 and 16 weeks post-dose).

The follow-up period (16 weeks) has been selected based on the predicted terminal half-life of AZD8233 in man (predicted to be 2 to 3 weeks), to cover at least 5 half-lives.

Following review of data from the study, the Safety Review Committee (SRC) may decide to:

* Adjust the window for sentinel dosing.
* Adjust the length of data collection prior to dose-escalation diction.
* Prolong the length of the stay at the Clinical Unit.
* Adjust the timing and number of assessments and/or blood/urine samples for subsequent cohorts.
* Adjust the length of the Follow-up Period. Each subject will be involved in the study for up to 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent before any study specific procedures.
2. Healthy male subjects aged 18 to 60 years (inclusive at Screening Visit) with suitable veins for cannulation or repeated venipuncture.
3. Have a body mass index (BMI) between 18 and 32 kg/m2 inclusive and weigh at least 60 kg and no more than 100 kg inclusive at the Screening Visit and Day -1.
4. Have a LDL-C ≥ 100 mg/dL < 190 mg/dL at the Screening Visit and Day -1, test may be repeated once for each visit at the discretion of the Investigator if out of the range.
5. Provision of signed, written and dated informed consent for optional genetic/biomarker research. If a subject declines to participate in the genetic component of the study, there will be no penalty or loss of benefit to the subject. The subject will not be excluded from other aspects of the study described in this protocol.

Exclusion Criteria:

1. History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. History or presence of GI, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
3. Any clinically important illness, medical/surgical procedure or trauma within 4weeks of the first administration of IMP.
4. Any laboratory values with the following deviations at the Screening Visit and/or Day -1, test may be repeated once for each visit at the discretion of the Investigator if out of range:

   4.1.Alanine aminotransferase (ALT)> upper limit of normal (ULN). 4.2.Aspartate aminotransferase (AST)> ULN. 4.3.Creatinine > ULN. 4.4.White blood cell (WBC)< LLN. 4.5.Hemoglobin< LLN. 4.6.Platelet count ≤150000/μL. 4.7.Activated partial thrombin time greater than ULN and PT greater than ULN. 4.8.Have an eGFR < 60mL/min. 4.9.Have an urinary albumin-to-creatinine ratio(ACR)> 3mg/μmol (30mg/g).
5. Any other clinically important abnormalities in clinical chemistry, hematology or urinalysis results, than those described under exclusion criterion number 4, as judged by the Investigator.
6. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody and human immunodeficiency virus (HIV).
7. Abnormal vital signs, after 10 minutes supine rest, with the following deviations at the Screening Visit and/or Day -1, test may be repeated once for each visit at the discretion of the Investigator if out of range:

   7.1.Systolic BP< 90mmHgor> 140mmHg. 7.2.Diastolic BP< 50mmHgor > 90mmHg. 7.3.Heart rate < 45 or > 85 beats per minute(bpm).
8. Any clinically important abnormalities in rhythm, conduction or morphology of the resting ECG and any clinically important abnormalities in the 12 Lead ECG as considered by the Investigator that may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology, particularly in the protocol defined primary lead or left ventricular hypertrophy at the Screening Visit or Day -1, test may be repeated once for each visit, at the discretion of the Investigator if out of range.

   8.1. Prolonged QTcF > 450 ms. 8.2. Shortened QTcF < 340 ms. 8.3. Family history of long QT syndrome. 8.4. PR (PQ) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation).

   8.5. PR (PQ) interval prolongation (> 240 ms) intermittent second (Wenckebach block while asleep is not exclusive) or third degree atrioventricular (AV) block, or AV dissociation.

   8.6. Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS > 110 ms. Subjects with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of e.g., ventricular hypertrophy or pre-excitation.
9. Known or suspected history of drug abuse as judged by the Investigator.
10. Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the previous 3 months before the Screening Visit.
11. History of alcohol abuse or excessive intake of alcohol as judged by the Investigator.
12. Positive screen for drugs of abuse, alcohol, or cotinine (nicotine) at the Screening Visit or positive screen for drugs of abuse or alcohol, on admission to the Clinical Unit.
13. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD8233.
14. Excessive intake of caffeine-containing drinks or food (e.g., coffee, tea, chocolate,) as judged by the Investigator.
15. Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks before the first administration of IMP.
16. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times t he recommended daily dose) and minerals during the 2 weeks before the first administration of IMP or longer if the medication has a long half-life.
17. Plasma donation within 1 month of the Screening Visit or any blood donation/blood loss > 500 mL during the 3 months before the Screening Visit.
18. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or 1 month after the last visit whichever is the longest. Note: subjects consented and screened, but not randomized in this study or a previous Phase 1 study, are not excluded.
19. Involvement of any Astra Zeneca or study site employee or their close relatives.
20. Judgment by the Investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the Screening Period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
21. Subjects who are vegans or have medical dietary restrictions.
22. Subjects who cannot communicate reliably with the Investigator.
23. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

    In addition, any of the following is regarded as a criterion for exclusion from the genetic research:
24. Previous bone marrow transplant.
25. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy male subjects with elevated LDL-C levels, aged 18 to 60 years that weigh at least 60 kg and no more than 100 kg inclusive.
Enrollment: 73 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2020-12-19 (Actual); Study Completion 2020-12-19 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) due to AZD8233 SC SAD treatment | From randomization to 4 months follow-up
  To assess AEs as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses. Serious AEs will be recorded from the time of informed consent.
Vital sign: Blood pressure [BP] | From screening to 4 month follow-up.
  To assess supine position systolic and diastolic BP as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses. Both SBP and DBP will be collected after the subject has rested in the supine position for at least 10 minutes.
Vital sign: Pulse rate | From screening to 4 month follow-up.
  To assess supine position pulse rate as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses. Pulse rate will be collected after the subject has rested in the supine position for at least 10 minutes.
Vital sign: Oral body temperature | From screening to 4 month follow-up.
  To assess oral body temperature as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses. Body temperature will be collected after the subject has rested in the supine position for at least 10 minutes.
Number of patients with abnormal findings in Resting 12-lead Electrocardiogram (ECG) | From screening to 4 month follow-up.
  To assess any clinically significant abnormalities in the cardiovascular system functioning using a 12-lead ECG as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses. ECG evaluations will be recorded after approximately 10 min resting in supine position.
Physical examination | From screening to 4 month follow-up.
  To assess physical examination as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses. Full (general appearance, skin, cardiovascular, respiratory, abdomen, head, and neck [including ears, eyes, nose, and throat], lymph nodes, thyroid, musculoskeletal and neurological systems) and brief (Abbreviated; general appearance, skin, cardiovascular system, respiratory and abdomen) physical examinations will be performed.
Laboratory assessments: Haematology - Blood cells count | From screening to 4 month follow-up.
  To assess red blood cells ( RBC) and white blood cells (WBC) count as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Haematology - Hemoglobin (Hb) | From screening to 4 month follow-up.
  To assess Hb as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Haematology - Haematocrit (HCT) | From screening to 4 month follow-up.
  To assess HCT (volume percentage of RBC in blod) as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Haematology - Mean corpuscular volume (MCV) | From screening to 4 month follow-up.
  To assess MCV as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Haematology - Mean corpuscular hemoglobin (MCH) | From screening to 4 month follow-up.
  To assess MCH as a variable of safety and tolerability following SC administration of single ascending doses.
Laboratory assessments: Haematology - Mean corpuscular hemoglobin concentration (MCHC) | From screening to 4 month follow-up.
  To assess MCHC as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Haematology - Differential count | From screening to 4 month follow-up.
  To assess differential WBC count absolute count of neutrophils, lymphocytes, monocytes, eosinophils and basophils as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Haematology - Platelets | From screening to 4 month follow-up.
  To assess platelets count as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Haematology - Reticulocytes absolute count | From screening to 4 month follow-up.
  To assess reticulocytes absolute count as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Serum clinical chemistry - Electrolytes | From screening to 4 month follow-up.
  To assess serum level of sodium, potassium, calcium and phosphate as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Serum clinical chemistry - Urea | From screening to 4 month follow-up.
  To assess serum level of urea as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Serum clinical chemistry - Creatinine | From screening to 4 month follow-up.
  To assess serum level of creatinine as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Serum clinical chemistry - Glucose (fasting) | From screening to 4 month follow-up.
  To assess serum fasting glucose level as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Serum clinical chemistry - Liver enzymes | From screening to 4 month follow-up.
  To assess serum of Alkaline phosphatase (ALP), Alanine aminotransferase (ALT), Aspartate aminotransferase (AST) and Gamma glutamyl transpeptidase (GGT) as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Serum clinical chemistry - Total Bilirubin | From screening to 4 month follow-up.
  To assess serum bilirubin (total) level as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Serum clinical chemistry - Cell enzymes | From screening to 4 month follow-up.
  To assess serum glutamate dehydrogenase and lactate dehydrogenase level as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Coagulation | From screening to 4 month follow-up.
  To assess activated partial thrombin time (aPTT) and prothrombin time (PT) as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Lipid Panel | From screening to 4 month follow-up.
  To assess serum level of high density lipoprotein, low density lipoprotein, triglycerides and total cholesterol as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Clinical Urinalysis - Glucose | From screening to 4 month follow-up.
  To assess urine glucose level as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Clinical Urinalysis - Protein | From screening to 4 month follow-up.
  To assess urine protein level as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Clinical Urinalysis - Blood | From screening to 4 month follow-up.
  To assess presence of blood in urine as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Clinical Urinalysis - Creatinine | From screening to 4 month follow-up.
  To assess urine creatinine level as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Clinical Urinalysis - Microscopy evaluation | From screening to 4 month follow-up.
  If protein or blood present in urine, levels of RBC, WBC, Casts (Cellular, Granular, Hyaline) will be assessed as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Renal Safety Biomarkers - Serum Creatinine | From screening to 4 month follow-up.
  To assess renal biomarker by evaluation of serum creatinine level, as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Renal Safety Biomarkers - Urine protein | From screening to 4 month follow-up.
  To assess renal biomarker by evaluation of urine protein level, as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Renal Safety Biomarkers - Estimated glomerular filtration rate (eGFR) | From screening to 4 month follow-up.
  To assess renal biomarker by evaluation of eGFR, as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Renal Safety Biomarkers -Urine Kidney Injury Molecule-1 (KIM-1) | From screening to 4 month follow-up.
  To assess renal biomarker by evaluation of urine KIM-1 level, as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Renal Safety Biomarkers - Urine Neutrophil gelatinase-associated lipocalin (NGAL) | From screening to 4 month follow-up.
  To assess renal biomarker by evaluation of NGAL level in urine, as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Renal Safety Biomarkers - Urine Alpha-glutathione S-transferase (Alpha-GST) | From screening to 4 month follow-up.
  To assess renal biomarker by evaluation of Alpha-GST level in urine, as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Immune Activation Response: High Sensitivity - C-reactive protein (hs-CRP) | Days 1 to 3 (pre-dose, 2, 4, 24 and 48 hours post-dose).
  To assess hs-CRP level as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Complement Activation panel | Day -1 and Days 1 to 3 (2, 4 and 24 hours post-dose).
  To assess chemotactic factors (C3a, C5a and Bp) levels as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Injection Site Reaction Examinations | At Days 1 to 4, week 1 to 14 and week 16.
  To assess injection site reactions in terms of size (mm), color (pale/light red/dark red) and itching (yes or no) as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Number of patients with abnormal findings in Telemetry | At Day -1 and Days 1 to 3 (Pre-dose to 24 hours post-dose)
  To assess heart rhythm and QRS pattern (heart conduction) as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses. ECG evaluations will be recorded after approximately 10 min resting in supine position.
Laboratory assessments: Serum clinical chemistry - Creatine kinase | From screening to 4 month follow-up.
  To assess serum level of creatine kinase as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Serum clinical chemistry - Bicarbonate | From screening to 4 month follow-up.
  To assess serum level of Bicarbonate as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Serum clinical chemistry - Direct bilirubin | From screening to 4 month follow-up.
  To assess serum level of direct bilirubin as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.
Laboratory assessments: Serum clinical chemistry -Uric acid | From screening to 4 month follow-up.
  To assess serum level of Uric acid as a variable of safety and tolerability of AZD8233 following SC administration of single ascending doses.

SECONDARY OUTCOMES:
Plasma PK analysis: Time delay between drug administration and the first observed concentration in plasma (tlag) | At treatment Days 1 to 3 (Pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose); Day 4 (72 hours post-dose); week 1 to 14 (1, 2, 4, 6, 8 and 12 weeks post-dose) and Final Follow-up Visit/ET Visit
  To characterize tlag of AZD8233 following SC administration of SAD.
Plasma PK analysis: Time to reach peak or maximum observed concentration following drug administration (tmax) | At treatment Days 1 to 3 (Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose); Day 4 (72 hours post-dose); week 1 to 14 (at 1, 2, 4, 6, 8 and 12 weeks post-dose) and Final Follow-up Visit/ET Visit
  To characterize tmax of AZD8233 following SC administration of SAD.
Plasma PK analysis: Maximum observed plasma concentration (Cmax) | At treatment Days 1 to 3 (Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose); Day 4 (72 hours post-dose); week 1 to 14 (at 1, 2, 4, 6, 8 and 12 weeks post-dose) and Final Follow-up Visit/ET Visit
  To characterize Cmax of AZD8233 following SC administration of SAD.
Plasma PK analysis: Area under the plasma concentration-curve from time zero to the time of last quantifiable analyte concentration (AUC[0-last]) | At treatment Days 1 to 3 (Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose); Day 4 (72 hours post-dose); week 1 to 14 (at 1, 2, 4, 6, 8 and 12 weeks post-dose) and Final Follow-up Visit/ET Visit
  To characterize AUC(0-last) of AZD8233 following SC administration of SAD.
Plasma PK analysis: Area under the concentration-time curve from time zero to 48 hours post-dose (AUC[0-48]) | At treatment Days 1 to 3 (Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose); Day 4 (72 hours post-dose); week 1 to 14 (at 1, 2, 4, 6, 8 and 12 weeks post-dose) and Final Follow-up Visit/ET Visit
  To characterize AUC(0-48) of AZD8233 following SC administration of SAD.
Plasma PK analysis: Area under the concentration-time curve from time zero extrapolated to infinity (AUC) | At treatment Days 1 to 3 (Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose); Day 4 (72 hours post-dose); week 1 to 14 (at 1, 2, 4, 6, 8 and 12 weeks post-dose) and Final Follow-up Visit/ET Visit
  To characterize AUC of AZD8233 following SC administration of SAD. AUC is estimated by AUC(0-last) + Clast/λz where Clast is the last observed quantifiable concentration.
Plasma PK analysis: Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | At treatment Days 1 to 3 (Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose); Day 4 (72 hours post-dose); week 1 to 14 (at 1, 2, 4, 6, 8 and 12 weeks post-dose) and Final Follow-up Visit/ET Visit
  To characterize CL/F of AZD8233 following SC administration of SAD.
Plasma PK analysis: Apparent volume of distribution for parent drug at terminal phase (extravascular administration) (Vz/F) | At treatment Days 1 to 3 (Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose); Day 4 (72 hours post-dose); week 1 to 14 (at 1, 2, 4, 6, 8 and 12 weeks post-dose) and Final Follow-up Visit/ET Visit
  To characterize Vz/F of AZD8233 following SC administration of SAD; estimated by dividing the apparent clearance (CL/F) by λz.
Plasma PK analysis: Half-life associated with the terminal slope (λz) of a semi-logarithmic concentration-time curve (t½z) | At treatment Days 1 to 3 (Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose); Day 4 (72 hours post-dose); week 1 to 14 (at 1, 2, 4, 6, 8 and 12 weeks post-dose) and Final Follow-up Visit/ET Visit
  To characterize t½z of AZD8233 following SC administration of SAD.
Plasma PK analysis: Mean Residence Time (MRT) | At treatment Days 1 to 3 (Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose); Day 4 (72 hours post-dose); week 1 to 14 (at 1, 2, 4, 6, 8 and 12 weeks post-dose) and Final Follow-up Visit/ET Visit
  To characterize MRT of AZD8233 following SC administration of SAD.
Urine PK analysis: Amount of analyte excreted unchanged in urine from time t1 to t2 (Ae[t1-t2]) | Treatment Days 1 to 3 (Pre-dose, 0-6, 6-12, 12-24, 24-36 and 36-48 hours post-dose)
  To characterize Ae(t1-t2) of AZD8233 following SC administration of SAD.
Urine PK analysis: Cumulative amount of analyte excreted at the last sampling interval (Ae[0-last]) | Treatment Days 1 to 3 (Pre-dose, 0-6, 6-12, 12-24, 24-36 and 36-48 hours post-dose)
  To characterize Ae(0-last) of AZD8233 following SC administration of SAD.
Urine PK analysis: Fraction of analyte excreted unchanged in urine from t1 to t2 (fe[t1-t2]) | Treatment Days 1 to 3 (Pre-dose, 0-6, 6-12, 12-24, 24-36 and 36-48 hours post-dose)
  To characterize fe(t1-t2) of AZD8233 following SC administration of SAD.
Urine PK analysis: Cumulative fraction of dose excreted unchanged into the urine from time zero to the last measured time-point for an analyte (fe[0-last]) | Treatment Days 1 to 3 (Pre-dose, 0-6, 6-12, 12-24, 24-36 and 36-48 hours post-dose)
  To characterize fe(0-last) of AZD8233 following SC administration of SAD; estimated by dividing Ae(0-last) by dose.
Urine PK analysis: Percentage of dose excreted unchanged into the urine from time zero to the last measured time-point for an analyte (%fe[0-last]) | Treatment Days 1 to 3 (Pre-dose, 0-6, 6-12, 12-24, 24-36 and 36-48 hours post-dose)
  To characterize %fe(0-last) of AZD8233 following SC administration of SAD; estimated by dividing Ae(0-last) by dose.
Urine PK analysis: Renal clearance of drug from plasma (CLR) | Treatment Days 1 to 3 (Pre-dose and then at 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose)
  To characterize CLR of AZD8233 following SC administration of SAD; estimated by dividing Ae(0-48) by AUC(0-48).
PD analysis: The effect of AZD8233 on cholesterol and related biomarkers | At screening, Day -1, Days 1 to 3 (pre-dose and 24 hours post-dose), Day 4 (72 hours post-dose), week 1 to 14 (at 1, 2, 3, 4, 6, 8, 10 and 12 weeks post-dose) and final follow-up visit/ET visit
  To assess the effect of AZD8233 on a PD variable (cholesterol and related biomarkers) following SC administration of single ascending doses. The results will be listed and summarized by treatment (dose level of AZD8233 or pooled placebo) including changes from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: David Han, M.D, Principal Investigator — PAREXEL Early Phase Clinical Unit-Los Angeles
Locations (1):
- Research Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home